CLINICAL TRIAL: NCT00708513
Title: Phase I/II Evaluation of Intraoperative Autotransfusion Filtration for Major Surgical Oncology Operations
Brief Title: Intraoperative Cell Saver Autotransfusion Use for Major Surgical Oncology Operations.
Acronym: Cellsaver
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, MD, University of Louisville
Other Study IDs: Cell Saver 704.03
Record Dates: First submitted 2008-06-27; First posted 2008-07-02 (Estimated); Last update posted 2013-10-21 (Estimated); Status verified 2013-10

CONDITIONS: Pancreaticoduodenectomy; Pancreatectomy; Esophagectomy; Gastrectomy; Hepatectomy
Keywords: Cell Saver; Liver Tumors; Liver Cancer; Surgical Oncology; Whipple; Blood Transfusion; Blood salvage; cancer surgery; blood loss
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to demonstrate the safety and benefit of auto-transfusion filtered blood in patients undergoing major surgical oncology procedures.

DETAILED DESCRIPTION:
Homologous blood transfusions during surgical procedures are becoming more challenging, due to lack of adequate reserves and the significant risks of transfusion reactions. Recent advances in the use of patient's own blood (autologous transfusion) has rapidly gained acceptance in major surgical procedures, however due to the requirement for prior planning and the expense of obtaining and storing a patient's blood prior to surgery this alternative is less than ideal.

This research study utilizes a third alternative, a technique called intraoperative autotransfusion, which successfully salvages a patient's blood during surgery and reinfuses the blood back into the patient. The blood salvaging device uses a filtration device that successfully filters out all tumor cells to prevent re-infusion of viable cancer cells.

This study is designed to demonstrate the safety and benefits of the blood salvaging device on patients undergoing major surgical oncology procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is undergoing a major surgical oncology procedure and has potential for extensive blood loss.
2. Subject is ≥ 18 years of age.
3. Subject or Subject's Legally Authorized Representative (LAR) has signed an IRB-approved informed consent form.

Exclusion Criteria:

1. Subject has medical, social, or psychological factors that, in the opinion of the Investigator, could impact safety or compliance with study procedures.
2. Subject is < 18 years of age.
3. Subject or Subject's LAR did not sign IRB-approved informed consent form.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical Oncology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2003-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of intra-operative ultrasound contrast (Definity) administration | Hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Robert CG Martin, MD, Principal Investigator — University of Louisville
Locations (2):
- United States (2):
  - Norton Healthcare, Louisville, Kentucky
  - University of Louisville Hospital, Louisville, Kentucky